CLINICAL TRIAL: NCT03027310
Title: Clinical and Physiological Studies of Tremor Syndromes
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170035; 17-N-0035
Record Dates: First submitted 2017-01-18; First posted 2017-01-23 (Estimated); Last update posted 2025-11-12 (Actual); Status verified 2025-11-07

CONDITIONS: Parkinson Disease; Dystonia; Essential Tremor
Keywords: Dystonic Tremor; Essential Tremor; Parkinsonism; Voice Tremor; Parkinson's Disease; Natural History
MeSH Terms: conditions — Parkinson Disease; Dystonia; Essential Tremor; Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: adult healthy volunteers
- tremor patients: adult patients with tremor

SUMMARY:
Background:

Researchers have some data on how the brain controls movement and why some people have tremor. But the causes of tremor are not fully known. Researchers want to study people with tremor to learn about changes in the brain and possible causes of tremor.

Objective:

To better understand how the brain controls movement, learn more about tremor, and train movement disorder specialists.

Eligibility:

People ages 18 and older with a diagnosed tremor syndrome

Healthy volunteers ages 18 and older

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Urine tests
* Clinical rating scales
* Health questions
* They may have electromyography (EMG) or accelerometry. Sensors or electrodes taped to the skin measure movement.

Participation lasts up to 1 year.

Some participants will have a visit to examine their tremor more. They may have rating scales, EMG, and drawing and writing tests.

Participants will be in 1 or more substudies. These will require up to 7 visits. Visits could include the following:

* EMG with accelerometry
* Small electrodes taped on the body give small electric shocks that stimulate nerves.
* MRI: Participants lie on a table that slides into a cylinder that takes pictures of the body while they do simple tasks.
* Small electrodes on the scalp record brain waves.
* A cone with detectors on the head measures brain activity while participants do tasks.
* A wire coil held on the scalp gives an electrical current that affects brain activity.
* Tests for thinking, memory, smell, hearing, or vision
* Electrodes on the head give a weak electrical current that affects brain activity.
* Photographs or videos of movement

Participant data may be shared with other researchers.

DETAILED DESCRIPTION:
Objectives

The purpose of this protocol is to study the phenotypic spectrum and the pathophysiology of tremor syndromes by performing small behavioral, electrophysiological and neuroimaging sub-studies. The protocol includes techniques with minimal risk (standard clinical evaluation, MRI, EEG, peripheral nerve stimulation, single and paired pulse TMS) and certain sub-studies may involve healthy volunteers. This protocol aims to study neurophysiological and behavioral outcomes in defined groups of patients with tremor syndromes, to inform future hypothesis-driven and confirmatory studies, which will be developed and submitted as separate protocols. For this purpose, we aim to conduct 1) pilot sub-studies, 2) individual patient investigations, 3) technical development studies.

Study population

We intend to enroll up to 300 patients with essential tremor and other isolated action tremor syndromes, as well as 150 healthy volunteers.

Design

This is a non-hypothesis driven study involving standardized phenotyping After patients and healthy volunteers complete a screening visit, patients will undergo a standardized phenotyping visit including clinical rating scales as well as electrophysiological tremorworkup. Patient and healthy controls may then be enrolled in sub-studies, and if a substudy leads to results of interest, a separate protocol will be submitted with a priori hypotheses, specific study design and power analysis adapted from the pilot or exploratory sub-studies performed in the present protocol.

Outcome measures

Outcome measures applied in this protocol involve methods for tremor phenotyping such as clinical rating scales and questionnaires, electrophysiological tremor studies, videotaped exam, as well as digitizing based tasks. During the sub-studies focused on the neurophysiological characterization of tremor syndromes, the following outcome measures will be applied: EMG: we will analyze tremor signals using spectral analyses, coherence analyses, and in combination with accelerometry, EEG, MEG, and TMS to explore tremor-networks. MRI: we will analyze measures such as the amplitude of the BOLD signal (fMRI); tractography between seed and target regions of interest (using DTI); morphometry of brain regions (using VBM); and different neurotransmitter levels in brain regions of interest (using MRS). EEG and MEG: we will quantify measures such as corticomuscular coherence, event- or task-related potentials, synchronization/desynchronization, and coherence between sensors or sources located close to the brain areas of interest. TMS: we will analyze measures such as MEP amplitude and central conduction time, as well as measures of cortical excitability and inhibition paradigms. Behavioral measures: we will quantify measures of voluntary movement involving tremor, reaction times to initiate movements, EMG patterns, movement kinematics (position, velocity, acceleration, curvature), eye movement. Actigraphy: We will quantify continuous recordings of motion sensors involving multiaxial accelerometers and gyroscopes. Furthermore, we may measure autonomic data during the course of experiments (such as blood pressure, skin co ductance, and respiratory rate) which would correlate to the outcome measures.

ELIGIBILITY:
* INCLUSION CRITERIA FOR TREMOR PATIENTS:
* Patients diagnosed with a tremor syndrome, including, but not limited to

  * Essential tremor (per definition of the Tremor Research Group)
  * Parkinson disease (per UK Brain Bank criteria)
  * Focal tremor such as isolated head tremor, voice tremor
  * Task-specific tremor such as primary writing tremor
  * Orthostatic tremor
  * Patients with other tremor syndromes such as dystonic tremor, intention tremor, etc.
* Age 18 or older
* Able to give informed consent
* Agree to not drink caffeine or alcohol for 12 hours before phenotyping and selected sub-study visits because both agents can modify brain activity and may confound outcome measures.

INCLUSION CRITERIA FOR HEALTHY VOLUNTEERS:

* Age 18 or older.
* Able to give informed consent.
* Agree to not consume caffeine or alcohol for 12 hours before selected sub-study visits because both agents may modify the activity of the brain during the study.

EXCLUSION CRITERIA FOR TREMOR PATIENTS:

* Problematic alcohol use, as defined by a score of 8 or higher on the WHO Alcohol Use Disorders Identification Test (AUDIT).
* History of a brain tumor, a stroke, traumatic brain injury, epilepsy or a history of seizures.
* History of psychotic disorder, Bipolar Disorder or a current depressive episode.
* History or clinical evidence of another neurologic disorder than a tremor syndrome as defined above, which may interfere with the ability to comply with protocol requirements or interpret the obtained results.

EXCLUSION CRITERIA FOR HEALTHY VOLUNTEERS:

* Have abnormal findings of clinical significance on the neurological examination that may affect the scientific integrity of the study
* Problematic alcohol use, as defined by a score of 8 or higher on the WHO Alcohol Use Disorders Identification Test (AUDIT)
* History of a brain tumor, a stroke, traumatic brain injury, epilepsy or a history of seizures.
* History of psychotic disorder, Bipolar Disorder or a current depressive episode.

ADDITIONAL EXCLUSION CRITERIA FOR MOVEMENT DISORDER PATIENTS AND HEALTHY VOLUNTEERS SPECIFICALLY FOR MRI:

We will follow the NMR Center guidelines for MR safety.

Some of the exclusions are:

* Have non-MRI compatible metal in the body, such as a cardiac pacemaker, brain stimulator, shrapnel, surgical metal, clips in the brain or on blood vessels, cochlear implants, artificial heart valves or ferromagnetic fragments in the eye or oral cavity as these make having an MRI unsafe.
* Unable to lie flat on the back for the expected length of the experiment.
* Have uncontrolled movements of the head.
* Have an abnormality on the brain imaging or neurologic examination not related to the diagnosis.
* Uncomfortable being in a small space for the expected length of the experiment.
* Non-removable body piercing or tattoo posing MRI risk
* Pregnancy.

ADDITIONAL EXCLUSION CRITERIA FOR TREMOR PATIENTS AND HEALTHY VOLUNTEERS FOR TMS AND MRI:

* Ferromagnetic metal in the cranial cavity or eye, e.g. aneurysm clip or ocular foreign body.
* Implanted electronic device including deep brain stimulation systems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Experimental subjects will include healthy volunteer subjects and patients with tremor syndromes including, but not limited to ET, PD-tremor, and dystonic tremor. The diagnosis will be made by a movement disorders neurologist at the NINDS movement disorders clinics. Healthy volunteers will be recruited for the following purposes: (1) to optimize data acquisition and analysis techniques; and (2) to serve as negative controls for clinical, imaging, and biological variables measured in the patient cohorts. Without data obtained from healthy volunteers, there is no way to determine whether subtle findings in tremor (e.g., physiological tremor) are truly abnormal. The inclusion of healthy volunteers therefore allows to correctly threshold and quantify observed abnormalities. Healthy volunteers may also include non-affected family members of patients with tremor
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
methods for tremor phenotyping | throughout protocol
  clinical rating scales and questionnaires, electrophysiological tremor studies, videotaped exam, as well as digitizing based tasks. EMG, EEG, MEG, TMS, MRI. Behavioral measures such as reaction times to initiate movements, EMG patterns, movement kinematics, eye movement.

CONTACTS AND LOCATIONS:
Overall Officials: Debra J Ehrlich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share all collected deidentified IPD at the request of others after publication. Data will not be sent until the applicable approvals and data sharing agreement has been obtained.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication.
Access Criteria: Requests will be considered on a case-by-case basis and we will try to uphold the NIH data-sharing directive. At the same time we may need IRB approval and/or data sharing agreements to be in place before we send data to others.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-N-0035.html